CLINICAL TRIAL: NCT06634368
Title: Pilot Study of Hospital GamePlan4Care for Family Caregivers of People With Dementia (CDA 21-143)
Brief Title: Pilot Study of Hospital GamePlan4Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CDX 24-003
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Caregivers
Keywords: Dementia; Hospitalization; Patient Discharge; Caregiver Burden
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: This is a single-blind, parallel group, randomized pilot trial of a 3-month caregiver support intervention for caregivers of hospitalized Veterans with dementia compared to health education. Participants will be assigned at random to the intervention (Hospital GamePlan4Care) or health education control. Assessment of the primary and secondary outcomes will occur pre-intervention at baseline and post-intervention at 1 and 3 months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hospital GamePlan4care (Experimental): Tailored caregiver skills training and support for caregiving for a person with dementia
  Interventions: Behavioral: Hospital GamePlan4Care
- Health Education (Active Comparator): Education on general caregiving topics.
  Interventions: Other: Health Education

INTERVENTIONS:
Behavioral: Hospital GamePlan4Care — The Hospital GamePlan4Care intervention will include access to a written VA Care Transitions handbook, access to the GamePlan4Care website for skills training, 11 emails encouraging them to visit the website, and four phone calls with a dementia care specialist to tailor the training to the caregiver's needs over a 3-month period.
  Arms: Hospital GamePlan4care
Other: Health Education — Caregivers in the health education arm will receive a VA Care Transitions Handbook, 4 emails with a weblink to a general caregiving topic, and 4 phone calls to confirm that the emails were received over a 3-month period.
  Arms: Health Education

SUMMARY:
Hospital stays are stressful for the family and friends who care for adults with dementia. Following hospital discharge, adults with dementia often have increased care needs, which places new caregiving demands on their family and friends. Family and friends are critical to ensuring that Veterans with dementia can live safely in the community following discharge. Healthcare systems have an opportunity to support family and friends of adults with dementia by addressing dementia-specific caregiving challenges that arise during the transition from hospital to home.

The investigators are comparing two different support programs for family and friends of hospitalized adults with dementia. The two programs are Hospital GamePlan4Care and Caregiver Education. Hospital GamePlan4Care was developed with feedback from people who care for Veterans with dementia. Hospital GamePlan4Care helps caregivers build skills to care for someone with dementia recently discharged from the hospital. It includes a written handbook, online training on the Hospital GamePlan4Care website, and phone calls with a dementia care specialist. The online training is tailored to the caregiver. The Caregiver Education program provides information that helps caregivers care for someone recently hospitalized. It includes a written handbook, recommendations for high-quality online resources, and phone calls with a dementia care specialist.

Both programs will start when the adult with dementia is hospitalized. Each program lasts at least three months. To be eligible, the caregiver must care for a Veteran with dementia admitted to the Michael E. DeBakey VA Medical Center in Houston, Texas. Caregivers interested in participating and passing eligibility screening will be enrolled in the study for at least three months. Each enrolled caregiver will have a 50% chance of being enrolled in the Hospital GamePlan4Care group or the Caregiver Education group (like flipping a coin). Both groups will be asked to complete several questionnaires about their needs as a caregiver and their well-being. Questionnaires will be completed at the beginning of the study and one and three months after the Veteran is discharged from the hospital. Each questionnaire should take 30-60 minutes to complete.

DETAILED DESCRIPTION:
The efficacy of support interventions designed for caregivers of adults with dementia and delivered as part of hospital care has not been established. Hospital GamePlan4Care is a new intervention that has been developed and tested with feedback from caregivers and health professionals. Hospital GamePlan4Care was feasible to implement during hospital care and acceptable to caregivers in a single-arm feasibility and acceptability pilot. There are no prior caregiver support interventions that include the same population (caregivers of adults with dementia), intervention delivery mechanism (web-based intervention), and practice setting (intervention started in the hospital and continued following discharge) to estimate effect sizes for a large randomized control trial of Hospital GamePlan4Care.This study will be a pilot single-blind randomized study comparing Hospital GamePlan4Care (intervention arm) to a Health Education Control arm (Caregiver Education). Caregivers will be assigned to the intervention or control arm in a ratio of 1:1. Each arm will continue for three months after the Veteran is discharged from the hospital.

Caregivers of adults with dementia will be recruited while the Veteran they care for is hospitalized. The research coordinator will complete the informed consent with the caregiver before the Veteran is discharged. All enrolled caregivers will receive a VA Care Transitions handbook. Following baseline data collection, enrolled caregivers will be randomized to Hospital GamePlan4Care or Caregiver Education arm in a 1:1 ratio using the randomization feature in VA REDCap. All Veterans and caregivers will receive standard hospital discharge planning and post-discharge care. A standard hospital discharge includes a consultation with an inpatient social worker or case manager, inpatient medication reconciliation, patient-centered written discharge instructions, a post-discharge phone call from the Veteran's primary care clinic, and scheduled follow-up appointments. The primary outcomes are caregiver-reported and will be measured 30 days and 90 days after hospital discharge.

Caregivers randomized to Hospital GamePlan4Care will receive 1) access to the Hospital GamePlan4Care website that includes training content relevant to caregivers during care transitions, such as learning how to complete new medical tasks, managing delirium, and addressing dementia behaviors, 2) 11 automated emails after hospital discharge that highlight Hospital GamePlan4Care training content and encourage caregivers to log into the website, and 3) four scheduled contacts with a Dementia Care Specialist after hospital discharge to tailor the intervention to the caregivers needs. Scheduled contacts with the Dementia Care Specialist will be on Day 2, Day 14, Day 28, and Day 60 after discharge.

Caregivers randomized to Caregiver Education will receive: 1) four automated emails after hospital discharge with recommended resources from the Home Alone Alliance, which provides high-quality training videos for caregivers, and 2) four scheduled phone calls with the Dementia Care Specialist after hospital discharge to confirm the emails were received and to see if the caregiver has any questions about the materials. Emails will be sent on Day 2, Day 14, Day 28, and Day 60 after discharge, and phone calls will be made after each email is sent.

The results from this study will inform the feasibility and sample size calculation for a multisite randomized controlled trial to test the efficacy of Hospital GP4C to improve caregiver-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* provide care for a Veteran with a diagnosis of Alzheimer's Disease or related dementias or a Veteran with a prescription for a medication for dementia listed in CPRS who is admitted to the hospital at the Michael E. DeBakey VA Medical Center
* Veteran must be experiencing signs of dementia as verified by a score of 2 or greater on the AD-8
* provide at least eight hours of care or supervision per week to the Veteran with dementia
* provide care primarily due to a personal relationship, rather than a financial relationship
* have access to a telephone
* have access to a tablet or computer with internet access
* report using the computer or tablet to access the internet at least three times per week
* speak English

Exclusion Criteria:

* unable to complete informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Zarit Caregiving Burden Interview (12-item) | Baseline, 30 days and 90 days
  Each item represents a statement related to an aspect of perceived burden. All questions are answered as never (0 points), rarely (1 point), sometimes (2 points), quite frequently (3 points), or nearly always (4 points). A total score will be obtained by summing all items with higher scores indicating higher rates of burden (range: 0-48).
Change in Center for Epidemiological Studies Depression Scale (CES-D) (10-item) | Baseline, 30 days, and 90 days
  The CES-D provides a list of feelings and behaviors. For each item, respondents report how often they have felt that way in the past week with each item receiving a score from 0-3. A total score will be obtained by summing scores for all items with higher scores indicating higher levels of depressed symptoms (range: 0-30).
Change in Self-Rated Health (1-item) | Baseline, 30 days, and 90 days
  The investigators will use the single self-rated health item: "In general, would you say your health is:" with response options of Excellent, Very Good, Good, Fair, and Poor
Change in Neuropsychiatric Inventory Questionnaire | Baseline, 30 days, and 90 days
  The Neuropsychiatric Inventory Questionnaire includes a list of 12 symptoms (e.g. delusions, hallucinations, agitation/aggression). For each symptom, the caregiver responds if the symptom was present in the past month (yes/no), the severity of the symptom if present (1-3), and the level of distress the caregiver feels due to that symptom (0-5). Higher scores indicate higher severity and greater distress due to that symptom.

SECONDARY OUTCOMES:
Change in Self-Efficacy for Caregiving (CSES-8) | Baseline, 30 days, and 90 days
  The CSES-8 asks questions about confidence in being able to manage different caregiving situations. Each question is rated on a 1 (not at all confident) to 10 (totally confident scale). The score of the scale is the mean of the eight items. Higher scores indicate greater self-efficacy.
Change in Benjamin Rose Institute Unmet Need Scale | Baseline, 30 days, and 90 days
  The Benjamin Rose Institute Unmet Need Scale includes 39 yes/no questions about different need that caregivers have (no=0, yes=1). The total score is a sum of all the yes responses. Higher scores indicate higher unmet needs.

OTHER OUTCOMES:
Change in VA Unplanned Acute Care Use | 30 days and 90 days
  Measure VA and VA-paid emergency room visits and unplanned readmissions.
Change in VA Home and Community-Based Services | 30 days and 90 days
  Measure VA and VA-paid Home and Community-Based Services, including home-based primary care, home skilled care, homemaker/home health aide, adult day health care, home hospice care, and respite care

CONTACTS AND LOCATIONS:
Overall Officials: Molly Horstman, MD MS, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide a de-identified dataset compliant with VA data security policy to the public upon request to the principal investigator.
Time Frame: After the data is analyzed and published